CLINICAL TRIAL: NCT06105463
Title: Response to Physical Activity in Women with Multiple Sclerosis Throughout the Menstrual Cycle (EMMA Project)
Brief Title: Multiple Sclerosis, Menstrual Cycle and Physical Acivity
Acronym: EMMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Jacobo Á. Rubio-Arias, Associate Professor, Universidad de Almeria
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: UALBIO2022/048; EXP_75066 (Other Grant/Funding Number: Consejo Superior de Deportes (Spain))
Record Dates: First submitted 2023-10-02; First posted 2023-10-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: strength training; High-Intensity Interval Training; Physical activity satisfaction; quality of life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: An randomized crossover trial and single-blind.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Women with Multiple Sclerosis (Experimental): Women diagnosed with Multiple Sclerosis by a certified neurologist
  Interventions: Other: Strength training sessions and High-interval intensity training sessions
- Women without Multiple Sclerosis (Active Comparator): Women not diagnosed with multiple sclerosis
  Interventions: Other: Strength training sessions and High-interval intensity training sessions

INTERVENTIONS:
Other: Strength training sessions and High-interval intensity training sessions — During strength training sessions, participants will perform 4 lower limb exercises, including bilateral leg press, unilateral leg extension, unilateral hip extension, and bilateral seated calf raise on conventional weight machines. The intensity of the session will be 70-75% of 1-RM, 4 sets, 10 repetitions (1-2 RIR) and 120 seconds rest between sets.
  During High-interval intensity training (HIIT) sessions, participants will perform 10 minutes of warm-up at 50% of peak power + 20 minutes of HIIT consisting of 30 seconds at 90% of peak power followed by 30 seconds of rest + 10 minutes of cool-down at 35-40% of peak power in cycloergometer.

SUMMARY:
This study aims to identify moderating variables that modify satisfaction with physical activity practice throughout the menstrual cycle (MC) in women with and without multiple sclerosis (MS) during High-Intensity Interval Training (HIIT) and strength training sessions, and to compare the acute effects of different types of physical activity sessions in women with and without MS. This study used a randomized crossover trial study and single-blind performed by women with MS, matched 1:1 based on age, lifestyle factors and country of residence, with women without MS to analyse the effect of physical activity practise on satisfaction, functionality, fatigue, and inflammatory profile throughout MC. Participants will visit the facilities approximately 10 times (4 preliminary familiarization visits and 6 visits to carry out a physical activity session in each phase of the MC) over a period of 3-4 months. Evaluation will comprise clinical, nutritional and psychological interviews including different variables such as satisfaction on physical activity; visual analogue scale of fatigue; abdominal obesity and anthropometric variables; dietary and nutritional monitoring; bioimpedance analysis; blood profile of hormone, inflammatory and cognitive function blood profile; neuromuscular strength, voluntary activation, and contractile properties; functional assessment (spasticity, knee angles, gait speed, walking endurance, balance, sit-to-stand test, timed up and go test); rating of perceived exertion; pain; muscle oxygen saturation; lactate; heart rate variability; quality of sleep and life; and body temperature. During the luteal phase, women with MS are expected to exhibit different acute responses to HIIT and strength training sessions compared to women without the disease.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 18-40 years;
* women with a menstrual cycle length of ≥ 21 days and ≤ 35 days of natural menstruation;
* absence of iron deficiency anaemia (serum ferritin > 20 μg/L, hemoglobin > 115 μg/L, transferrin saturation > 16%)
* being in a stable phase of the disease,
* to ambulate autonomously for more than 100 meters

Exclusion Criteria:

* a score < 2 or > 6 on the Expanded Disability Status Scale (EDSS);
* experienced a relapse in the 12 months prior to enrolment;
* received corticosteroid treatment in the previous 2 months;
* participated in a structured exercise programme in the past 6 months;
* secondary amenorrhoea (absence of ≥ 3 consecutive periods despite not being pregnant and having previous menstruation);
* used or currently use hormonal contraceptives for 3 months before recruitment
* reported musculoskeletal or neurological injuries not associated with MS, recent surgical interventions, or pregnancies in the previous year,
* have unrelated diseases to MS

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-06 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with physical activity | Before sessions (strength and High-interval intensity training session)
  Satisfaction with physical activity will be assessed using an eight-item scale adapted from previous studies. The questionnaire begins with the statement "When I am doing physical activity" followed by the items "I am satisfied with the results of/I am satisfied with/I enjoy/I feel good when I have done/I notice positive results if I have done physical activity," "Physical activity has many advantages," and "I find physical activity nice/difficult." Responses to this single-item question will be measured on a 5-point scale, ranging from 1 (very dissatisfied) to 5 (very satisfied). Satisfaction will be assessed before, immediately following the training session, and at 24, 48, and 72 hours.
Satisfaction with physical activity | Immediately after sessions (strength and High-interval intensity training session)
  Satisfaction with physical activity will be assessed using an eight-item scale adapted from previous studies. The questionnaire begins with the statement "When I am doing physical activity" followed by the items "I am satisfied with the results of/I am satisfied with/I enjoy/I feel good when I have done/I notice positive results if I have done physical activity," "Physical activity has many advantages," and "I find physical activity nice/difficult." Responses to this single-item question will be measured on a 5-point scale, ranging from 1 (very dissatisfied) to 5 (very satisfied). Satisfaction will be assessed before, immediately following the training session, and at 24, 48, and 72 hours.
Satisfaction with physical activity | 24 hours after sessions (strength and High-interval intensity training session)
  Satisfaction with physical activity will be assessed using an eight-item scale adapted from previous studies. The questionnaire begins with the statement "When I am doing physical activity" followed by the items "I am satisfied with the results of/I am satisfied with/I enjoy/I feel good when I have done/I notice positive results if I have done physical activity," "Physical activity has many advantages," and "I find physical activity nice/difficult." Responses to this single-item question will be measured on a 5-point scale, ranging from 1 (very dissatisfied) to 5 (very satisfied). Satisfaction will be assessed before, immediately following the training session, and at 24, 48, and 72 hours.
Satisfaction with physical activity | 48 hours after sessions (strength and High-interval intensity training session)
  Satisfaction with physical activity will be assessed using an eight-item scale adapted from previous studies. The questionnaire begins with the statement "When I am doing physical activity" followed by the items "I am satisfied with the results of/I am satisfied with/I enjoy/I feel good when I have done/I notice positive results if I have done physical activity," "Physical activity has many advantages," and "I find physical activity nice/difficult." Responses to this single-item question will be measured on a 5-point scale, ranging from 1 (very dissatisfied) to 5 (very satisfied). Satisfaction will be assessed before, immediately following the training session, and at 24, 48, and 72 hours.
Satisfaction with physical activity | 72 hours after sessions (strength and High-interval intensity training session)
  Satisfaction with physical activity will be assessed using an eight-item scale adapted from previous studies. The questionnaire begins with the statement "When I am doing physical activity" followed by the items "I am satisfied with the results of/I am satisfied with/I enjoy/I feel good when I have done/I notice positive results if I have done physical activity," "Physical activity has many advantages," and "I find physical activity nice/difficult." Responses to this single-item question will be measured on a 5-point scale, ranging from 1 (very dissatisfied) to 5 (very satisfied). Satisfaction will be assessed before, immediately following the training session, and at 24, 48, and 72 hours.
Visual analog scale of fatigue (VAS-F) | Before sessions (strength and High-interval intensity training session)
  This scale is subdivided into two subscales: fatigue and energy. The VAS-F presents a horizontal line measuring 100mm in length, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line that corresponds to their perception of fatigue severity between these two endpoints. The fatigue subscale is organized starting from the most positive items to the most negative ones. Conversely, the energy subscale ranges from the most negative to the most positive items. A high score on the VAS-F indicates a low score on the energy subscale and a high level of severity on the fatigue subscale. This scale is widely used both in the general population and in clinical patients due to its brevity, ease of use, and comprehensibility.
Visual analog scale of fatigue (VAS-F) | Immediately after sessions (strength and High-interval intensity training session)
  This scale is subdivided into two subscales: fatigue and energy. The VAS-F presents a horizontal line measuring 100mm in length, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line that corresponds to their perception of fatigue severity between these two endpoints. The fatigue subscale is organized starting from the most positive items to the most negative ones. Conversely, the energy subscale ranges from the most negative to the most positive items. A high score on the VAS-F indicates a low score on the energy subscale and a high level of severity on the fatigue subscale. This scale is widely used both in the general population and in clinical patients due to its brevity, ease of use, and comprehensibility.
Visual analog scale of fatigue (VAS-F) | 24 hours after sessions (strength and High-interval intensity training session)
  This scale is subdivided into two subscales: fatigue and energy. The VAS-F presents a horizontal line measuring 100mm in length, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line that corresponds to their perception of fatigue severity between these two endpoints. The fatigue subscale is organized starting from the most positive items to the most negative ones. Conversely, the energy subscale ranges from the most negative to the most positive items. A high score on the VAS-F indicates a low score on the energy subscale and a high level of severity on the fatigue subscale. This scale is widely used both in the general population and in clinical patients due to its brevity, ease of use, and comprehensibility.
Visual analog scale of fatigue (VAS-F) | 48 hours after sessions (strength and High-interval intensity training session)
  This scale is subdivided into two subscales: fatigue and energy. The VAS-F presents a horizontal line measuring 100mm in length, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line that corresponds to their perception of fatigue severity between these two endpoints. The fatigue subscale is organized starting from the most positive items to the most negative ones. Conversely, the energy subscale ranges from the most negative to the most positive items. A high score on the VAS-F indicates a low score on the energy subscale and a high level of severity on the fatigue subscale. This scale is widely used both in the general population and in clinical patients due to its brevity, ease of use, and comprehensibility.
Visual analog scale of fatigue (VAS-F) | 72 hours after sessions (strength and High-interval intensity training session)
  This scale is subdivided into two subscales: fatigue and energy. The VAS-F presents a horizontal line measuring 100mm in length, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line that corresponds to their perception of fatigue severity between these two endpoints. The fatigue subscale is organized starting from the most positive items to the most negative ones. Conversely, the energy subscale ranges from the most negative to the most positive items. A high score on the VAS-F indicates a low score on the energy subscale and a high level of severity on the fatigue subscale. This scale is widely used both in the general population and in clinical patients due to its brevity, ease of use, and comprehensibility.

SECONDARY OUTCOMES:
Subjective Sleep Quality Questionnaire | Before sessions (strength and High-interval intensity training session)
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnarie. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (awakened much too early [1] - did not wake up early [3]), e) ease of awakening (very difficult [1] - very easy [5]), f) feeling of restfulness (did not rest at all [1] - completely rested [3]), and g) sleep sufficiency (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | Immediately after sessions (strength and High-interval intensity training session)
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnarie. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (awakened much too early [1] - did not wake up early [3]), e) ease of awakening (very difficult [1] - very easy [5]), f) feeling of restfulness (did not rest at all [1] - completely rested [3]), and g) sleep sufficiency (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | 24 hours after sessions (strength and High-interval intensity training session)
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnarie. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (awakened much too early [1] - did not wake up early [3]), e) ease of awakening (very difficult [1] - very easy [5]), f) feeling of restfulness (did not rest at all [1] - completely rested [3]), and g) sleep sufficiency (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | 48 hours after sessions (strength and High-interval intensity training session)
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnarie. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (awakened much too early [1] - did not wake up early [3]), e) ease of awakening (very difficult [1] - very easy [5]), f) feeling of restfulness (did not rest at all [1] - completely rested [3]), and g) sleep sufficiency (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | 72 hours after sessions (strength and High-interval intensity training session)
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnarie. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (awakened much too early [1] - did not wake up early [3]), e) ease of awakening (very difficult [1] - very easy [5]), f) feeling of restfulness (did not rest at all [1] - completely rested [3]), and g) sleep sufficiency (no, definitely too little [1] - yes, definitely enough [5]).
Sleep Quality Measured by Actigraphy | Before sessions (strength and High-interval intensity training session)
  Actigraphy-based sleep quality will be assessed using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK). This device employs a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower threshold of actigraphic sensitivity will be set at 80 counts/epoch. The Actiwatch sleep analysis software will be utilized. Data analysis will begin at the start of the nocturnal rest (bedtime) and conclude at the beginning of daytime activity (wake time). Sleep efficiency (%), percentage of time spent asleep, time in bed (minutes), actual sleep time (minutes), actual wake time (minutes), number of awakenings, and average duration of each awakening (minutes) will be measured
Sleep Quality Measured by Actigraphy | Immediately after sessions (strength and High-interval intensity training session)
  Actigraphy-based sleep quality will be assessed using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK). This device employs a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower threshold of actigraphic sensitivity will be set at 80 counts/epoch. The Actiwatch sleep analysis software will be utilized. Data analysis will begin at the start of the nocturnal rest (bedtime) and conclude at the beginning of daytime activity (wake time). Sleep efficiency (%), percentage of time spent asleep, time in bed (minutes), actual sleep time (minutes), actual wake time (minutes), number of awakenings, and average duration of each awakening (minutes) will be measured
Sleep Quality Measured by Actigraphy | 24 hours after sessions (strength and High-interval intensity training session)
  Actigraphy-based sleep quality will be assessed using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK). This device employs a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower threshold of actigraphic sensitivity will be set at 80 counts/epoch. The Actiwatch sleep analysis software will be utilized. Data analysis will begin at the start of the nocturnal rest (bedtime) and conclude at the beginning of daytime activity (wake time). Sleep efficiency (%), percentage of time spent asleep, time in bed (minutes), actual sleep time (minutes), actual wake time (minutes), number of awakenings, and average duration of each awakening (minutes) will be measured
Sleep Quality Measured by Actigraphy | 48 hours after sessions (strength and High-interval intensity training session)
  Actigraphy-based sleep quality will be assessed using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK). This device employs a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower threshold of actigraphic sensitivity will be set at 80 counts/epoch. The Actiwatch sleep analysis software will be utilized. Data analysis will begin at the start of the nocturnal rest (bedtime) and conclude at the beginning of daytime activity (wake time). Sleep efficiency (%), percentage of time spent asleep, time in bed (minutes), actual sleep time (minutes), actual wake time (minutes), number of awakenings, and average duration of each awakening (minutes) will be measured
Sleep Quality Measured by Actigraphy | 72 hours after sessions (strength and High-interval intensity training session)
  Actigraphy-based sleep quality will be assessed using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK). This device employs a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower threshold of actigraphic sensitivity will be set at 80 counts/epoch. The Actiwatch sleep analysis software will be utilized. Data analysis will begin at the start of the nocturnal rest (bedtime) and conclude at the beginning of daytime activity (wake time). Sleep efficiency (%), percentage of time spent asleep, time in bed (minutes), actual sleep time (minutes), actual wake time (minutes), number of awakenings, and average duration of each awakening (minutes) will be measured
Heart Rate Variability | Before sessions (strength and High-interval intensity training session)
  Heart rate variability (HRV) measurements will be taken using a Polar H10 heart rate sensor to record heartbeats during sleep. Analysis of HRV variables will be conducted using Kubios HRV software. Poincaré plot, time-domain, and frequency-domain analyses will be performed. Analysed time-domain variables include:: mean heart rate, mean R-R interval, standard deviation of consecutive R-R intervals, square root of the mean squared differences of successive R-R intervals, and the proportion of consecutive intervals differing by more than 50 ms. Fast Fourier Transform (FFT) will be employed to calculate frequency-domain spectral components. High-frequency (HF; 0.15-1.0 Hz) and low-frequency (LF; 0.04-0.15 Hz) power components will be computed as integrals of their respective power spectral density curves.
Heart Rate Variability | Immediately after sessions (strength and High-interval intensity training session)
  Heart rate variability (HRV) measurements will be taken using a Polar H10 heart rate sensor to record heartbeats during sleep. Analysis of HRV variables will be conducted using Kubios HRV software. Poincaré plot, time-domain, and frequency-domain analyses will be performed. Analysed time-domain variables include:: mean heart rate, mean R-R interval, standard deviation of consecutive R-R intervals, square root of the mean squared differences of successive R-R intervals, and the proportion of consecutive intervals differing by more than 50 ms. Fast Fourier Transform (FFT) will be employed to calculate frequency-domain spectral components. High-frequency (HF; 0.15-1.0 Hz) and low-frequency (LF; 0.04-0.15 Hz) power components will be computed as integrals of their respective power spectral density curves.
Heart Rate Variability | 24 hours after sessions (strength and High-interval intensity training session)
  Heart rate variability (HRV) measurements will be taken using a Polar H10 heart rate sensor to record heartbeats during sleep. Analysis of HRV variables will be conducted using Kubios HRV software. Poincaré plot, time-domain, and frequency-domain analyses will be performed. Analysed time-domain variables include:: mean heart rate, mean R-R interval, standard deviation of consecutive R-R intervals, square root of the mean squared differences of successive R-R intervals, and the proportion of consecutive intervals differing by more than 50 ms. Fast Fourier Transform (FFT) will be employed to calculate frequency-domain spectral components. High-frequency (HF; 0.15-1.0 Hz) and low-frequency (LF; 0.04-0.15 Hz) power components will be computed as integrals of their respective power spectral density curves.
Heart Rate Variability | 48 hours after sessions (strength and High-interval intensity training session)
  Heart rate variability (HRV) measurements will be taken using a Polar H10 heart rate sensor to record heartbeats during sleep. Analysis of HRV variables will be conducted using Kubios HRV software. Poincaré plot, time-domain, and frequency-domain analyses will be performed. Analysed time-domain variables include:: mean heart rate, mean R-R interval, standard deviation of consecutive R-R intervals, square root of the mean squared differences of successive R-R intervals, and the proportion of consecutive intervals differing by more than 50 ms. Fast Fourier Transform (FFT) will be employed to calculate frequency-domain spectral components. High-frequency (HF; 0.15-1.0 Hz) and low-frequency (LF; 0.04-0.15 Hz) power components will be computed as integrals of their respective power spectral density curves.
Heart Rate Variability | 72 hours after sessions (strength and High-interval intensity training session)
  Heart rate variability (HRV) measurements will be taken using a Polar H10 heart rate sensor to record heartbeats during sleep. Analysis of HRV variables will be conducted using Kubios HRV software. Poincaré plot, time-domain, and frequency-domain analyses will be performed. Analysed time-domain variables include:: mean heart rate, mean R-R interval, standard deviation of consecutive R-R intervals, square root of the mean squared differences of successive R-R intervals, and the proportion of consecutive intervals differing by more than 50 ms. Fast Fourier Transform (FFT) will be employed to calculate frequency-domain spectral components. High-frequency (HF; 0.15-1.0 Hz) and low-frequency (LF; 0.04-0.15 Hz) power components will be computed as integrals of their respective power spectral density curves.
Heart Rate Variability | During sessions (strength and High-interval intensity training session)
  Heart rate variability (HRV) measurements will be taken using a Polar H10 heart rate sensor to record heartbeats during sleep. Analysis of HRV variables will be conducted using Kubios HRV software. Poincaré plot, time-domain, and frequency-domain analyses will be performed. Analysed time-domain variables include:: mean heart rate, mean R-R interval, standard deviation of consecutive R-R intervals, square root of the mean squared differences of successive R-R intervals, and the proportion of consecutive intervals differing by more than 50 ms. Fast Fourier Transform (FFT) will be employed to calculate frequency-domain spectral components. High-frequency (HF; 0.15-1.0 Hz) and low-frequency (LF; 0.04-0.15 Hz) power components will be computed as integrals of their respective power spectral density curves.
Muscle oxygen saturation | During sessions (strength and High-interval intensity training session)
  SMO2 of the right and left lateral quadriceps will be measured during sessions using a near-infrared spectroscopy system, the Moxy 3-Sensor Bundle (Fortiori Design LLC, Hutchinson, MN, USA). The average SMO2 will be calculated throughout the entire training session on both legs simultaneously.
Lactate | During sessions (strength and High-interval intensity training session)
  A portable lactate analyser (Lactate Scout system, RedMed, Warsaw, Poland) which measures lactate concentration using the principle of enzymatic determination by photometric reflection will be used. During the exercise sessions, capillary blood samples from the will be collected 1) at basal level (before the protocol and warm-up); 2) 1 min post-session (1 min after the end of the last high-intensity bout), 3) 3 min post-session and 4) 30 min post-session.
Maximum oxygen consumption | During sessions (strength and High-interval intensity training session)
  The maximum oxygen consumption achieved during an incremental test to exhaustion shall be measured using an ergo-spirometer.
Body composition | Before sessions (strength and High-interval intensity training session)
  Bioimpedance analysis: 100 μA (1 KHz) and 500 μA (5, 5, 50, 250, 500, and 1000 kHz), and a 100-240 V
Body composition | Immediately after sessions (strength and High-interval intensity training session)
  Bioimpedance analysis: 100 μA (1 KHz) and 500 μA (5, 5, 50, 250, 500, and 1000 kHz), and a 100-240 V
Hormonal profile | Before sessions (strength and High-interval intensity training session)
  To determine and monitor sexual function according to the menstrual cycle hormone criteria, serum hormone concentrations will be analysed, and 17β-estradiol, progesterone, prolactin, LH, FSH, TSH and testosterone 23 before each training session.
Hormonal profile | Immediately after sessions (strength and High-interval intensity training session)
  To determine and monitor sexual function according to the menstrual cycle hormone criteria, serum hormone concentrations will be analysed, and 17β-estradiol, progesterone, prolactin, LH, FSH, TSH and testosterone 23 before each training session.
Inflammatory profile | Before sessions (strength and High-interval intensity training session)
  IFN-γ as a marker associated with the pathogenesis of the disease, IL-6, TNF-α as pro-inflammatory markers and IL-10, β1 (TGF-b1) as anti-inflammatory markers will be assessed. All these markers shall be assessed before and at 30 and 60 minutes immediately after the session.
Inflammatory profile | Immediately after sessions (strength and High-interval intensity training session)
  IFN-γ as a marker associated with the pathogenesis of the disease, IL-6, TNF-α as pro-inflammatory markers and IL-10, β1 (TGF-b1) as anti-inflammatory markers will be assessed. All these markers shall be assessed before and at 30 and 60 minutes immediately after the session.
Cognitive function | Before sessions (strength and High-interval intensity training session)
  Brain-derived neurotrophic factor (BDNF) is a member of the neurotrophin family, several studies have found associations between exercise, circulating levels of BDNF, hippocampal volume, and cognitive function in the general population 74 and neurodegenerative disorders.
Cognitive function | Immediately after sessions (strength and High-interval intensity training session)
  Brain-derived neurotrophic factor (BDNF) is a member of the neurotrophin family, several studies have found associations between exercise, circulating levels of BDNF, hippocampal volume, and cognitive function in the general population 74 and neurodegenerative disorders.
Rate of force development | Before sessions (strength and High-interval intensity training session)
  the participants will be seated in a chair, with both legs flexed at a 90 degree angle and the ankle of the tested firmly strapped to a customised device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). Subsequently, participants will be instructed to apply "as much force as possible, as fast as possible" on each trial. Participants will perform three maximal contractions of two seconds each, with a rest of three minutes between contractions.RFD and the time at which the value is observed will be analysed in the following ranges: 0-50 ms: RFDearly, 0-200 ms: RFDlate and peak slope: RFDpeak. The right leg will be tested first, and the repetition in which the highest peak value of each leg is observed will be analysed.
Rate of force development | Immediately after sessions (strength and High-interval intensity training session)
  the participants will be seated in a chair, with both legs flexed at a 90 degree angle and the ankle of the tested firmly strapped to a customised device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). Subsequently, participants will be instructed to apply "as much force as possible, as fast as possible" on each trial. Participants will perform three maximal contractions of two seconds each, with a rest of three minutes between contractions. RFD and the time at which the value is observed will be analysed in the following ranges: 0-50 ms: RFDearly, 0-200 ms: RFDlate and peak slope: RFDpeak. The right leg will be tested first, and the repetition in which the highest peak value of each leg is observed will be analysed.
Maximal Voluntary Activation | Before sessions (strength and High-interval intensity training session)
  the participants will be seated in a chair, with both legs flexed at a 90 degree angle and the ankle of the tested firmly strapped to a customised device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). Subsequently, participants will be instructed to apply "as much force as possible, as fast as possible" on each trial. Participants will perform three maximal contractions of two seconds each, with a rest of three minutes between contractions.
Maximal Voluntary Activation | Immediately after sessions (strength and High-interval intensity training session)
  the participants will be seated in a chair, with both legs flexed at a 90 degree angle and the ankle of the tested firmly strapped to a customised device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). Subsequently, participants will be instructed to apply "as much force as possible, as fast as possible" on each trial. Participants will perform three maximal contractions of two seconds each, with a rest of three minutes between contractions.
Contractile properties of muscle | Before sessions (strength and High-interval intensity training session)
  To measure neural drive, sEMG activity of the vastus lateralis of the right leg will be recorded during the MVIC. The preparation of the skin will involve shaving, abrasion, and cleansing with alcohol. Following SENIAM Guidelines, the upper electrode of each pair (Ambu Blue Sensor SP, Ambu A/S, Denmark) will be placed over the largest part of the vastus lateralis. Transparent paper will be used to map exact electrode placements for subsequent measurements. EMG activity will be analysed using the following time intervals: 0-50 ms (EMG 0 to 50), 0 to 200 ms (EMG 0 to 200), peak of EMG and EMG time-to-peak. The EMG peak during MVIC will represent maximal neural drive.
Contractile properties of muscle | Immediately after sessions (strength and High-interval intensity training session)
  To measure neural drive, sEMG activity of the vastus lateralis of the right leg will be recorded during the MVIC. The preparation of the skin will involve shaving, abrasion, and cleansing with alcohol. Following SENIAM Guidelines, the upper electrode of each pair (Ambu Blue Sensor SP, Ambu A/S, Denmark) will be placed over the largest part of the vastus lateralis. Transparent paper will be used to map exact electrode placements for subsequent measurements. EMG activity will be analysed using the following time intervals: 0-50 ms (EMG 0 to 50), 0 to 200 ms (EMG 0 to 200), peak of EMG and EMG time-to-peak. The EMG peak during MVIC will represent maximal neural drive.
Central activation ratio | Before sessions (strength and High-interval intensity training session)
  Two bipolar stimulating electrodes (10 × 15 cm) will be positioned and secured on the proximal and distal portions of the quadriceps of the right leg. Signal 6.0 software (CED, Cambridge, England) will control the electrical stimulation characteristics, which will be 100 Hz, 50 pulses, length 0.009 s, and interval 0.01 s. The stimulus intensity will be established at 40-50% of MVIC
Central activation ratio | Immediately after sessions (strength and High-interval intensity training session)
  Two bipolar stimulating electrodes (10 × 15 cm) will be positioned and secured on the proximal and distal portions of the quadriceps of the right leg. Signal 6.0 software (CED, Cambridge, England) will control the electrical stimulation characteristics, which will be 100 Hz, 50 pulses, length 0.009 s, and interval 0.01 s. The stimulus intensity will be established at 40-50% of MVIC
Maximal upper limb strength | Before sessions (strength and High-interval intensity training session)
  ): Participants will stand with their elbows fully extended and separated from the trunk. In this position, isometric handgrip strength will be measured for 5 seconds using the electronic hand dynamometer (TL-LSC100, Trailite, Ahaus, Germany). Participants will perform three trials in each hand (right and left), and a rest interval of 60 seconds will be given between attempts. The highest value achieved will be recorded.
Maximal upper limb strength | Immediately after sessions (strength and High-interval intensity training session)
  ): Participants will stand with their elbows fully extended and separated from the trunk. In this position, isometric handgrip strength will be measured for 5 seconds using the electronic hand dynamometer (TL-LSC100, Trailite, Ahaus, Germany). Participants will perform three trials in each hand (right and left), and a rest interval of 60 seconds will be given between attempts. The highest value achieved will be recorded.
Spasticity | Before sessions (strength and High-interval intensity training session)
  The pendulum test will be used for spasticity assessment. Metrics including the relaxation index (RI), the count of oscillations, duration of oscillations, and the extent of the first swing excursion will be computed.
Spasticity | Immediately after sessions (strength and High-interval intensity training session)
  The pendulum test will be used for spasticity assessment. Metrics including the relaxation index (RI), the count of oscillations, duration of oscillations, and the extent of the first swing excursion will be computed.
Gait speed | Before sessions (strength and High-interval intensity training session)
  Gait speed will be measured using the 10-meter walk test (10-MWT), where 2 photocells (Ergotest Technology AS, Langesund, Norway) will be placed at 6 and 10 meters to record the time. Participants will perform the test as fast as possible without running, completing it twice with a 2-minute rest in between. Participants will be consistently encouraged throughout the 10-MWT. The recorded time for the slowest walking trial (in seconds) will be utilized for analysis
Gait speed | Immediately after sessions (strength and High-interval intensity training session)
  Gait speed will be measured using the 10-meter walk test (10-MWT), where 2 photocells (Ergotest Technology AS, Langesund, Norway) will be placed at 6 and 10 meters to record the time. Participants will perform the test as fast as possible without running, completing it twice with a 2-minute rest in between. Participants will be consistently encouraged throughout the 10-MWT. The recorded time for the slowest walking trial (in seconds) will be utilized for analysis
Balance | Before sessions (strength and High-interval intensity training session)
  during the static balance measurements, participants will stand quietly on a portable force platform (Ergotest Technology AS, Langesund, Norway) while being barefoot, maintaining a shoulder-width stance, and letting their arms hang at their sides. Each participant will perform two trials lasting 30 seconds each, with both eyes open, and another two trials of the same duration with their eyes closed.
Balance | Immediately after sessions (strength and High-interval intensity training session)
  during the static balance measurements, participants will stand quietly on a portable force platform (Ergotest Technology AS, Langesund, Norway) while being barefoot, maintaining a shoulder-width stance, and letting their arms hang at their sides. Each participant will perform two trials lasting 30 seconds each, with both eyes open, and another two trials of the same duration with their eyes closed.
Sit-to-Stand Test (STS) | Before sessions (strength and High-interval intensity training session)
  Participants will be positioned in an upright manner on an adjustable chair (considering lower limb length; 90º knee flexion) with arms crossed over the chest. They will be instructed to rise to a standing position as swiftly as possible. Video recording with iphone 14 will be employed to determine the conclusion of the movement when both the participant's trunk and knees are fully extended. This test will be conducted twice, and the most successful trial will be utilized for analysis.
Sit-to-Stand Test (STS) | Immediately after sessions (strength and High-interval intensity training session)
  Participants will be positioned in an upright manner on an adjustable chair (considering lower limb length; 90º knee flexion) with arms crossed over the chest. They will be instructed to rise to a standing position as swiftly as possible. Video recording with iphone 14 will be employed to determine the conclusion of the movement when both the participant's trunk and knees are fully extended. This test will be conducted twice, and the most successful trial will be utilized for analysis.
Timed Up and Go Test (TUG) | Before sessions (strength and High-interval intensity training session)
  In a prompt manner, participants will transition from a seated to a standing position. They will then walk a distance of 3 meters forward, execute a turn, walk back, and resume the seated posture. This test will be repeated twice. A video recording will be used to ascertain the fastest time among the two trials, which will subsequently be used for analysis
Timed Up and Go Test (TUG) | Immediately after sessions (strength and High-interval intensity training session)
  In a prompt manner, participants will transition from a seated to a standing position. They will then walk a distance of 3 meters forward, execute a turn, walk back, and resume the seated posture. This test will be repeated twice. A video recording will be used to ascertain the fastest time among the two trials, which will subsequently be used for analysis
Rating of Perceived Exertion (RPE) | Before sessions (strength and High-interval intensity training session)
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each of the proposed exercises within the session), and after the training session using the Borg 6-20 RPE
Rating of Perceived Exertion (RPE) | Immediately after sessions (strength and High-interval intensity training session)
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each of the proposed exercises within the session), and after the training session using the Borg 6-20 RPE
Delayed-Onset Muscle Soreness (DOMS) | Before sessions (strength and High-interval intensity training session)
  a 10-point Likert scale will be employed to evaluate pain, where 1 = no pain and 10 = unbearable pain.
Delayed-Onset Muscle Soreness (DOMS) | Immediately after sessions (strength and High-interval intensity training session)
  a 10-point Likert scale will be employed to evaluate pain, where 1 = no pain and 10 = unbearable pain.
Muscle pain sensitivity | Before sessions (strength and High-interval intensity training session)
  an algometer FPIX (Wagner's instruments, USA) will be used to quantify pain sensitivity in specific muscle regions (same anatomical areas where spasticity is measured). The algometer will be calibrated according to the manufacturer's guidelines. Participants will be instructed to indicate their initial pain threshold. The rounded tip of the algometer will ensure an even application of pressure
Muscle pain sensitivity | Immediately after sessions (strength and High-interval intensity training session)
  an algometer FPIX (Wagner's instruments, USA) will be used to quantify pain sensitivity in specific muscle regions (same anatomical areas where spasticity is measured). The algometer will be calibrated according to the manufacturer's guidelines. Participants will be instructed to indicate their initial pain threshold. The rounded tip of the algometer will ensure an even application of pressure
Fat mass | Baseline Measurements
  The percentage of body fat (%) and the kilograms of fat mass (kg) of the participants will be obtained using the ISAK method of anthropometric profiling.
Muscle mass | Baseline Measurements
  The percentage of muscle mass (%) and the kilograms of muscle mass (kg) of the participants will be obtained using the ISAK method of anthropometric profiling.
Bone mass | Baseline Measurements
  The percentage of bone mass (%) and the kilograms of bone mass (kg) of the participants will be obtained using the ISAK method of anthropometric profiling.
Dietary and nutritional monitoring | Baseline Measurements
  Following the outlined schedule for dietary assessment, participants will be guided through the core elements of the "Dietary and Nutritional Monitoring Protocol."
Physical activity levels | Baseline measurements
  The International Physical Activity Questionnaire (IPAQ) will be administered. The telephone short version consisting of 7 items will be utilized. This version provides information about the time spent on performing moderate and vigorous-intensity activities, time dedicated to walking, and time spent sitting during a workday. It is designed for use with young people and adults aged 15-69 years. Physical activity will be recorded in METs (Metabolic Equivalent of Task or METs Units)
Physical activity levels | 7 days after the end of the study
  The International Physical Activity Questionnaire (IPAQ) will be administered. The telephone short version consisting of 7 items will be utilized. This version provides information about the time spent on performing moderate and vigorous-intensity activities, time dedicated to walking, and time spent sitting during a workday. It is designed for use with young people and adults aged 15-69 years. Physical activity will be recorded in METs (Metabolic Equivalent of Task or METs Units)
Walking endurance | Baseline measurements
  Participants will undergo the 6-minute walk test (6-MWT), during which they will walk at their self-selected preferred speed to assess walking endurance. The testing track will be rectangular, with corners marked by cones. Participants will be allowed to rest during the test if needed, but the time will not pause during these resting periods. The total distance covered (in meters) will be recorded. An investigator will be present during the test to accompany the participants, though no conversation will occur. This test will only be performed during baseline evaluations.
Physical self-perception | Through study completion, an average of 3 times per month, up to 10 weeks.
  The evaluation of physical self-perception will comprise six subscales aimed at gauging self-perception in various dimensions, including sports competence, physical condition, attractive body, physical strength, general physical self-perception, and general self-perception. Participants' responses will be organized using a 5-point Likert scale, with each subscale score having the potential to span from 6 to 36 points. A higher score will indicate a positive physical self-perception.
Catastrophizing Pain Scale | Through study completion, an average of 3 times per month, up to 10 weeks.
  The Catastrophizing Pain Scale will be used to assess feelings of catastrophizing related to pain (such as painful experiences). Subscale scores encompassing rumination and helplessness will be examined. Each of the 13 questions will be rated on a 5-point scale, with the endpoints ranging from <0> "not at all" to <4> "all the time." A lower score will indicate minimal or no pain catastrophizing.
Modified Fatigue Impact Scale (MFIS) | Through study completion, an average of 3 times per month, up to 10 weeks.
  The perception of fatigue will be measured using the MFIS, this scale is a 21-item multidimensional questionnaire that assesses the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84).
Multiple Sclerosis Quality of Life-54 (MSQoL-54) | Through study completion, an average of 3 times per month, up to 10 weeks.
  Participants will be filled out the Multiple Sclerosis Quality of Life-54 (MSQoL-54) questionnaire. The MSQoL-54 is a structured, self-report questionnaire comprising 14 sub-scales: physical function, physical role limitations, emotional role limitations, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, sexual function, satisfaction with sexual function, change in health, and overall quality of life. Two summary scores, the physical health composite summary and the mental health composite summary, can be derived from the MSQoL-54 questionnaire. Elevated scores in each subscale or summary score will indicate an improved quality of life.
State anxiety and trait anxiety (STAI) | Through study completion, an average of 3 times per month, up to 10 weeks.
  The STAI will be used to measure state and trait anxiety. This questionnaire assesses and discriminates the temporary psychological state in a given situation (state anxiety; 20 items), as well as the more stable character trait of attitudes and temperaments (trait anxiety; 20 items). This questionnaire is especially useful for the diagnosis of anxiety problems in non-psychiatric patients. It is based on a 4-point Likert scale, with a range of scores on each subscale from 10 to 40 points. A higher score on each of the subscales reflects higher state or trait anxiety, respectively.
Body temperature | Through study completion, an average of 3 times per month, up to 10 weeks.
  To capture thermal images, a PIR UC 605 thermographic camera (Infratec, Barcelona, Spain) will be used, equipped with an impressive infrared resolution of 640 x 480 pixels and an impressive thermal sensitivity of less than 0.06 ºC. Calibration of the camera will be conducted according to the manufacturer's recommendations, as well as recommendations from previous studies. The camera will be connected at least 30 min prior to all evaluations to allow stabilisation of its thermal sensor.
  Three measurements shall be performed following the Glamorgan protocol, designed to provide accurate measurements of body thermography

CONTACTS AND LOCATIONS:
Locations (1):
- University of Almeria, Almería, Almeria, Spain

REFERENCES:
- [Derived] Rubio-Arias JA, Ramos-Campo DJ, Romero-Parra N, Andreu-Caravaca L, Martinez-Rodriguez A, Esteban-Garcia P, Lopez-Liria R, Molina-Torres G, Ventura-Miranda MI, Martos-Bonilla A, Rando-Martin A, Carrasco-Poyatos M, Alacid F, Ferrer-Contreras MDC, Cupeiro R. Response to physical activity of females with multiple sclerosis throughout the menstrual cycle: a protocol for a randomised crossover trial (EMMA Project). BMJ Open Sport Exerc Med. 2023 Nov 21;9(4):e001797. doi: 10.1136/bmjsem-2023-001797. eCollection 2023. PMID 38022757